CLINICAL TRIAL: NCT04305106
Title: The Efficacy and Safety of Bevacizumab in Patients With Severe Covid-19: a Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Trial
Brief Title: Bevacizumab in Patients With Severe Covid-19
Acronym: BEST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: China-Japan Friendship Hospital (Other); Renmin Hospital of Wuhan University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Zhejing Provincial People's Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Anqing Municipal Hospital (Other); First Affiliated Hospital of Wannan Medical College (Other); The Fourth Affiliated Hospital Zhejing University School of Medicine (Unknown); Shandong Provincial Hospital (Other Government); Linyi People's Hospital (Other); Jining Medical University (Other); Jining First People's Hospital (Other); Weifang Second People's Hospital (Unknown); Weifang Medical University (Other); Yantai Yuhuangding Hospital (Other); Weihai Municipal Hospital (Other); Rizhao People's Hospital (Other); Qingdao Municipal Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Weifang People's Hospital (Other); Weifang Hospital of Traditional Chinese Medicine (Unknown); Zibo Central Hospital (Other Government); Zibo Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLEmer
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Bevacizumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab (Experimental): Bevacizumab 7.5mg/kg body weight, intravenous drip, single-dose administration, and standard of care, including prophylactic doses of low molecular weight heparin or unfractionated heparin without contraindications, and therapeutic doses of anticoagulants with the evidence of thrombosis risk or occurrence.
  Interventions: Drug: Bevacizumab; Other: Standard care
- Placebo (Placebo Comparator): Placebo (inactive excipient) 7.5mg/kg body weight, intravenous drip, single-dose administration, and standard of care, including prophylactic doses of low molecular weight heparin or unfractionated heparin without contraindications, and therapeutic doses of anticoagulants with the evidence of thrombosis risk or occurrence.
  Interventions: Other: Placebo; Other: Standard care

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (7.5mg/kg BW) + Saline (100ml) Bevacizumab will be administered in a single dose with no less than 90 minutes of intravenous infusion under ECG monitoring.
  Other Names: Recombinant anti-VEGF humanized monoclonal antibody injection
  Arms: Bevacizumab
Other: Placebo — Placebo (7.5mg/kg BW) + Saline (100ml) The placebo drug will be administered in a single dose with no less than 90 minutes of intravenous infusion under ECG monitoring.
  Other Names: Inactive excipient
  Arms: Placebo
Other: Standard care — Standard care, including prophylactic doses of low molecular weight heparin or unfractionated heparin without contraindications, and therapeutic doses of anticoagulants with the evidence of thrombosis risk or occurrence.

SUMMARY:
The novel coronavirus (SARS-CoV-2) is a new strain of coronavirus found in human in 2019, which causes epidemic worldwide. Novel coronavirus disease (COVID-19) causes acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) in patients with severe COVID-19. Pulmonary edema is the key detrimental feature of ALI/ARDS. Autopsy of patients died from COVID-19 reported that, pulmonary mucus exudation was more severe and obvious than SARS infection. Pulmonary CT scanning and pathological findings also suggest that pulmonary edema caused by inflammatory exudation is a distinguished feature of COVID-19. Vascular endothelial growth factor (VEGF), also known as vascular permeability factor (VPF), is known as the most potent factor to increase vascular permeability, with the induction effect 50,000 times stronger than histamine. Bevacizumab is an anti-VEGF recombinant humanized monoclonal antibody, which has been used in anti-tumor treatment since 2004, with considerable reliability and clinical safety. This trial will provide high level evidence to answer whether bevacizumab is efficacy and safe medication for patients with severe COVID-19.

DETAILED DESCRIPTION:
Evident increase of VEGF levels in serum has been displayed on novel pneumonia patients. The investigators also conducted a pilot study of 93 patients with severe COVID-19 that confirmed the significantly elevated level of plasma and serum VEGF.

At the beginning of 2020, the investigators proposed the concept of using anti-VEGF treatment for patients with severe COVID-19 and conducted a pilot study (NCT04275414). Among the 27 enrolled participants treated with bevacizumab, it was found that the clinical recovery status, PaO2/FiO2, and pulmonary exudation on imaging were significantly improved than the external controls in the same center during the same period. This provides good preliminary basis for this RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, both genders;
2. Confirmed COVID-19 diagnosis (any body fluid tested positive for SARS-CoV-2 nucleic acid by PCR, or positive for SARS-CoV-2 antigen);
3. Respiratory rate ≥ 30 times/min, partial pressure of oxygen (PaO2)/ fraction of inspiration O2 (FiO2)≤ 300mmHg (1mmHg = 0.133kPa), or SpO2 ≤ 93% at rest without supplemental oxygen;
4. Article (3) above is newly appeared within 7 days;
5. Chest radiography or computed tomography shows bilateral chest infiltrates.

Exclusion Criteria:

1. Unable to obtain informed consent.
2. Physician with more than 5 years of clinical experience determines that death was inevitable within 24 hours.
3. Severe hepatic dysfunction (Child Pugh score ≥ C, or AST> 5 times the upper limit); Severe renal dysfunction (estimated glomerular filtration rate ≤ 30mL/ min/1.73 m2) or receive continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
4. Uncontrolled hypertension (sitting systolic blood pressure> 160mmHg, or diastolic blood pressure>100mmHg); previous history of hypertension crisis or hypertensive encephalopathy.
5. Poorly controlled heart diseases, such as NYHA class II and above cardiac insufficiency, unstable angina pectoris, myocardial infarction within 1 year before enrollment, supraventricular or ventricular arrhythmia need treatment or intervention.
6. Severe or above chronic obstructive pulmonary disease (GOLD grade, FEV1/FVC < 0.5).
7. Hereditary bleeding tendency or coagulopathy;
8. Arterial/venous thromboembolic events within 6 months before enrollment, such as ischemic stroke, transient ischemic attack, deep venous thrombosis, pulmonary embolism, etc. Severe vascular disease (including aneurysms or arterial thrombosis requiring surgery) within 6 months before enrollment.
9. Unhealed wounds, active gastric ulcers or fractures. Gastrointestinal perforation, gastrointestinal fistula, abdominal abscess, visceral fistula formation within 6 months before enrollment. Major surgery (including preoperative Chest biopsy) or major trauma (such as a fracture) within 28 days before enrollment. May have surgery during the trial.
10. Severe, active bleeding such as hemoptysis, gastrointestinal bleeding, central nervous system bleeding, and nosebleeds within 1 month before enrollment.
11. Malignant tumors within 5 years before enrollment.
12. Allergic to bevacizumab or its components.
13. Active tuberculosis, uncontrollable infection, untreated active hepatitis or HIV-positive patients.
14. Pregnant and lactating women and those planning to get pregnant.
15. Participated in other clinical trials, not considered suitable for this study by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The time from randomization to clinical improvement | 28 days
  The time from randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale or live discharge from the hospital, whichever comes first.

SECONDARY OUTCOMES:
Intubation rate | From date of randomization until the date of discharge, up to 28 days
  Intubation rate
Duration of mechanical ventilation (days) | From date of randomization until the date of discharge, up to 28 days
  Days of mechanical ventilation
Duration of non-invasive ventilator or nasal high flow oxygen inhalation | From date of randomization until the date of discharge, up to 28 days
  Days of non-invasive ventilator or nasal high flow oxygen inhalation
All-cause mortality | From date of randomization until the date of discharge, up to 60 days
  All-cause mortality
Time to reach level 1 on the seven-category ordinal scale | up to 60 days
  Days from randomization to the clinical status of reaching level 1 on the seven--category ordinal scale
PaO2/FiO2 level | day 1, day 3, day 7 and day 14 after randomization, or before discharge
  The ratio of partial pressure of oxygen to fraction of inspiration O2
Improvement of pulmonary lesions | day 7 and day 14 after randomization, or before discharge
  The change of volumes of pulmonary exudation shown on CT compared to baseline
Improvement of lymphocyte count | day 7 and day 14 after randomization, or before discharge
  The change of the level of lymphocyte count compared to baseline
Improvement of CRP | day 7 and day 14 after randomization, or before discharge
  The change of the level of C-reactive protein compared to baseline
Improvement of LDH | day 7 and day 14 after randomization, or before discharge
  The change of the level of lactate dehydrogenase compared to baseline
SAE, AE | From date of randomization until the date of discharge, up to 28 days
  Serious adverse event, adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Yihai Cao, Dr, Principal Investigator — Qilu Hospital of Shandong University, Karolinska Institutet; Yuguo Chen, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
We will share the study protocol, SAP, ICF, CSR and analytic code on the day of article publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: On the day of article publication.
Access Criteria: By inquiring of principal investigator or central contact person.

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Pang J, Xu F, Aondio G, Li Y, Fumagalli A, Lu M, Valmadre G, Wei J, Bian Y, Canesi M, Damiani G, Zhang Y, Yu D, Chen J, Ji X, Sui W, Wang B, Wu S, Kovacs A, Revera M, Wang H, Jing X, Zhang Y, Chen Y, Cao Y. Efficacy and tolerability of bevacizumab in patients with severe Covid-19. Nat Commun. 2021 Feb 5;12(1):814. doi: 10.1038/s41467-021-21085-8. PMID 33547300